CLINICAL TRIAL: NCT00798161
Title: A Phase III Randomised, Double-blind, Placebo-controlled Parallel Group Study to Compare the Efficacy and Safety of Twice Daily Administration of the Free Combination of BI 1356 2.5 mg + Metformin 500 mg, or of BI 1356 2.5 mg + Metformin 1000 mg, With the Individual Components of Metformin (500 mg or 1000 mg Twice Daily), and BI 1356 (5.0 mg Once Daily) Over 24 Weeks in Drug Naive or Previously Treated (4 Weeks Wash-out and 2 Weeks Placebo run-in) Type 2 Diabetic Patients With Insufficient Glycaemic Control
Brief Title: Safety and Efficacy of Linagliptin (BI 1356) Plus Metformin in Type 2 Diabetes, Factorial Design
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1218.46; 2008-001640-40 (EudraCT Number: EudraCT)
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Results first posted 2011-08-04 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2013-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin; Metformin

ARMS (6):
- BI 1356 + metformin (Experimental): BI 1356 low dose + metformin 500 mg, twice daily
  Interventions: Drug: BI 1356 + metformin
- matching placebo (Placebo Comparator): matching placebo
  Interventions: Drug: matching placebo
- BI 1356+ Metformin (Experimental): BI 1356 low dose + metformin 1000 mg, twice daily
  Interventions: Drug: Bi 1356 + metformin
- Metformin (Active Comparator): Metformin 500 mg, twice daily
  Interventions: Drug: Metformin
- metformin (Active Comparator): Metformin 1000 mg, twice daily
  Interventions: Drug: metformin
- BI 1356 (Experimental): BI 1356 high dose, once daily
  Interventions: Drug: BI 1356

INTERVENTIONS:
Drug: BI 1356 — BI 1356 high dose tablet, once daily
  Arms: BI 1356
Drug: BI 1356 + metformin — BI 1356 low dose tablet + Metformin 500 mg tablet, twice daily
  Arms: BI 1356 + metformin
Drug: Bi 1356 + metformin — BI 1356 low dose tablet + Metformin 1000 mg tablet, twice daily
  Arms: BI 1356+ Metformin
Drug: Metformin — Metformin 500 mg tablet, twice daily
  Arms: Metformin
Drug: metformin — metformin 1000 mg tablet, twice daily
  Arms: metformin
Drug: matching placebo — matching placebo
  Arms: matching placebo

SUMMARY:
The objective of the randomised part of the study is to investigate the efficacy and safety of BI 1356 plus metformin compared to BI 1356 or metformin alone given for 24 weeks to drug naive or previously treated (4 weeks wash-out, 2 weeks placebo run-in) type 2 diabetic patients with insufficient glycaemic control. For the open-label part of the study the objective is to estimate the efficacy and safety of BI 1356 and metformin in type 2 diabetic patients with very poor glycaemic control for 24 weeks

ELIGIBILITY:
Inclusion criteria:

Patients with type 2 diabetes (drug naive or pre-treated) with insufficient glycaemic control (HbA1c higher or equal than 7.5 to less than 11.0 %), with very poor glycaemic control (HbA1c higher or equal than 11.0 %) who are not eligible for randomisation to be included in the open-label arm

Exclusion criteria:

Myocardial infarction, stroke or transient ischemic attack (TIA), unstable or acute congestive heart failure, impaired hepatic function, treatment with rosiglitazone or pioglitazone, with a GLP1 analogue, with insulin, with anti-obesity drugs, with systemic steroids, renal failure or impairment, gastric bypass

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 857 (Actual)
Dates: Start 2008-12; Primary Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (138):
- Canada (9):
  - 1218.46.11005 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 1218.46.11003 Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - 1218.46.11002 Boehringer Ingelheim Investigational Site, Red Deer, Alberta
  - 1218.46.11006 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1218.46.11008 Boehringer Ingelheim Investigational Site, Winnipeg, Manitoba
  - 1218.46.11004 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1218.46.11007 Boehringer Ingelheim Investigational Site, Oakville, Ontario
  - 1218.46.11009 Boehringer Ingelheim Investigational Site, Oshawa, Ontario
  - 1218.46.11010 Boehringer Ingelheim Investigational Site, Toronto, Ontario
- Croatia (6):
  - 1218.46.38502 Boehringer Ingelheim Investigational Site, Karlovac
  - 1218.46.38503 Boehringer Ingelheim Investigational Site, Krapinske Toplice
  - 1218.46.38504 Boehringer Ingelheim Investigational Site, Osijek
  - 1218.46.38505 Boehringer Ingelheim Investigational Site, Rijeka
  - 1218.46.38501 Boehringer Ingelheim Investigational Site, Sisak
  - 1218.46.38506 Boehringer Ingelheim Investigational Site, Zagreb
- Estonia (3):
  - 1218.46.37202 Boehringer Ingelheim Investigational Site, Pärnu
  - 1218.46.37201 Boehringer Ingelheim Investigational Site, Tallinn
  - 1218.46.37203 Boehringer Ingelheim Investigational Site, Tallinn
- France (41):
  - 1218.46.3303D Boehringer Ingelheim Investigational Site, Aire Sur l'Aadour
  - 1218.46.3308B Boehringer Ingelheim Investigational Site, Bischheim
  - 1218.46.3305A Boehringer Ingelheim Investigational Site, Bourges
  - 1218.46.3304F Boehringer Ingelheim Investigational Site, Bousse
  - 1218.46.3306D Boehringer Ingelheim Investigational Site, Carresse-Cassaber
  - 1218.46.3308C Boehringer Ingelheim Investigational Site, Gambsheim
  - 1218.46.3305D Boehringer Ingelheim Investigational Site, Garchizy
  - 1218.46.3301A Boehringer Ingelheim Investigational Site, Grenoble Cédex
  - 1218.46.3305B Boehringer Ingelheim Investigational Site, Guérigny
  - 1218.46.3304A Boehringer Ingelheim Investigational Site, Jarny
  - 1218.46.3302D Boehringer Ingelheim Investigational Site, La Riche
  - 1218.46.3307A Boehringer Ingelheim Investigational Site, La Seyne-sur-Mer
  - 1218.46.3307E Boehringer Ingelheim Investigational Site, La Seyne-sur-Mer
  - 1218.46.3305G Boehringer Ingelheim Investigational Site, Lury-sur-Arnon
  - 1218.46.3304D Boehringer Ingelheim Investigational Site, Mars-la-Tour
  - 1218.46.3304B Boehringer Ingelheim Investigational Site, Mondelange
  - 1218.46.3303A Boehringer Ingelheim Investigational Site, Mont-de-Marsan
  - 1218.46.3303C Boehringer Ingelheim Investigational Site, Mont-de-Marsan
  - 1218.46.3303E Boehringer Ingelheim Investigational Site, Mont-de-Marsan
  - 1218.46.3304C Boehringer Ingelheim Investigational Site, Moûtiers
  - 1218.46.3308F Boehringer Ingelheim Investigational Site, Mundolsheim
  - 1218.46.3305C Boehringer Ingelheim Investigational Site, Nevers
  - 1218.46.3305E Boehringer Ingelheim Investigational Site, Nevers
  - 1218.46.3306A Boehringer Ingelheim Investigational Site, Orthez
  - 1218.46.3306C Boehringer Ingelheim Investigational Site, Orthez
  - 1218.46.3306E Boehringer Ingelheim Investigational Site, Orthez
  - 1218.46.3306F Boehringer Ingelheim Investigational Site, Orthez
  - 1218.46.3304E Boehringer Ingelheim Investigational Site, Pont-à-Mousson
  - 1218.46.3302B Boehringer Ingelheim Investigational Site, Saint-Avertin
  - 1218.46.3302C Boehringer Ingelheim Investigational Site, Saint-Avertin
  - 1218.46.3303B Boehringer Ingelheim Investigational Site, Saint-Martin-d'Oney
  - 1218.46.3306B Boehringer Ingelheim Investigational Site, Salies-de-Béarn
  - 1218.46.3302E Boehringer Ingelheim Investigational Site, Savonnières
  - 1218.46.3308A Boehringer Ingelheim Investigational Site, Strasbourg
  - 1218.46.3308D Boehringer Ingelheim Investigational Site, Strasbourg
  - 1218.46.3308E Boehringer Ingelheim Investigational Site, Strasbourg
  - 1218.46.3307B Boehringer Ingelheim Investigational Site, Toulon
  - 1218.46.3307C Boehringer Ingelheim Investigational Site, Toulon
  - 1218.46.3307D Boehringer Ingelheim Investigational Site, Toulon
  - 1218.46.3302A Boehringer Ingelheim Investigational Site, Tours
  - 1218.46.3304H Boehringer Ingelheim Investigational Site, Vandœuvre-lès-Nancy
- Germany (6):
  - 1218.46.49002 Boehringer Ingelheim Investigational Site, Bad Dürrheim-Sunthausen
  - 1218.46.49001 Boehringer Ingelheim Investigational Site, Bad Mergentheim
  - 1218.46.49006 Boehringer Ingelheim Investigational Site, Cologne
  - 1218.46.49003 Boehringer Ingelheim Investigational Site, München
  - 1218.46.49008 Boehringer Ingelheim Investigational Site, Neuwied
  - 1218.46.49007 Boehringer Ingelheim Investigational Site, Schauenburg
- India (19):
  - 1218.46.91009 Boehringer Ingelheim Investigational Site, Aurangabad
  - 1218.46.91007 Boehringer Ingelheim Investigational Site, Babgalore
  - 1218.46.91001 Boehringer Ingelheim Investigational Site, Bangalore
  - 1218.46.91004 Boehringer Ingelheim Investigational Site, Bangalore
  - 1218.46.91012 Boehringer Ingelheim Investigational Site, Bangalore
  - 1218.46.91011 Boehringer Ingelheim Investigational Site, Bhopal
  - 1218.46.91003 Boehringer Ingelheim Investigational Site, Chennai
  - 1218.46.91020 Boehringer Ingelheim Investigational Site, Chennai
  - 1218.46.91018 Boehringer Ingelheim Investigational Site, Hyderadad
  - 1218.46.91008 Boehringer Ingelheim Investigational Site, Jaipur
  - 1218.46.91019 Boehringer Ingelheim Investigational Site, Madurai
  - 1218.46.91013 Boehringer Ingelheim Investigational Site, Maharashtra
  - 1218.46.91002 Boehringer Ingelheim Investigational Site, Manipal
  - 1218.46.91015 Boehringer Ingelheim Investigational Site, Mumbai
  - 1218.46.91014 Boehringer Ingelheim Investigational Site, Nagpur
  - 1218.46.91017 Boehringer Ingelheim Investigational Site, New Delhi
  - 1218.46.91016 Boehringer Ingelheim Investigational Site, P.O Trivandrum
  - 1218.46.91010 Boehringer Ingelheim Investigational Site, Pune
  - 1218.46.91006 Boehringer Ingelheim Investigational Site, West Bengal
- Lithuania (3):
  - 1218.46.37001 Boehringer Ingelheim Investigational Site, Kaunas
  - 1218.46.37004 Boehringer Ingelheim Investigational Site, Kaunas
  - 1218.46.37003 Boehringer Ingelheim Investigational Site, Vilnius
- Mexico (9):
  - 1218.46.52006 Boehringer Ingelheim Investigational Site, Aguascalientes
  - 1218.46.52002 Boehringer Ingelheim Investigational Site, Cuernavaca
  - 1218.46.52003 Boehringer Ingelheim Investigational Site, Guadalajara
  - 1218.46.52004 Boehringer Ingelheim Investigational Site, Guadalajara
  - 1218.46.52007 Boehringer Ingelheim Investigational Site, México
  - 1218.46.52008 Boehringer Ingelheim Investigational Site, México
  - 1218.46.52001 Boehringer Ingelheim Investigational Site, Pachuca
  - 1218.46.52010 Boehringer Ingelheim Investigational Site, Tijuana
  - 1218.46.52009 Boehringer Ingelheim Investigational Site, Veracruz
- Netherlands (13):
  - 1218.46.31004 Boehringer Ingelheim Investigational Site, 's-Hertogenbosch
  - 1218.46.31005 Boehringer Ingelheim Investigational Site, 's-Hertogenbosch
  - 1218.46.31001 Boehringer Ingelheim Investigational Site, Almere Stad
  - 1218.46.31008 Boehringer Ingelheim Investigational Site, Beek
  - 1218.46.31002 Boehringer Ingelheim Investigational Site, Beek en Donk
  - 1218.46.31010 Boehringer Ingelheim Investigational Site, Breda
  - 1218.46.31011 Boehringer Ingelheim Investigational Site, Eindhoven
  - 1218.46.31013 Boehringer Ingelheim Investigational Site, Groningen
  - 1218.46.31012 Boehringer Ingelheim Investigational Site, Leiderdrop
  - 1218.46.31016 Boehringer Ingelheim Investigational Site, Nijmegen
  - 1218.46.31009 Boehringer Ingelheim Investigational Site, Rotterdam
  - 1218.46.31014 Boehringer Ingelheim Investigational Site, Velp
  - 1218.46.31015 Boehringer Ingelheim Investigational Site, Zoetermeer
- Romania (5):
  - 1218.46.40001 Boehringer Ingelheim Investigational Site, Alba Iulia
  - 1218.46.40005 Boehringer Ingelheim Investigational Site, Galati
  - 1218.46.40003 Boehringer Ingelheim Investigational Site, Oradea
  - 1218.46.40002 Boehringer Ingelheim Investigational Site, Ploieşti
  - 1218.46.40004 Boehringer Ingelheim Investigational Site, Satu Mare
- Russia (8):
  - 1218.46.70001 Boehringer Ingelheim Investigational Site, Moscow
  - 1218.46.70002 Boehringer Ingelheim Investigational Site, Moscow
  - 1218.46.70003 Boehringer Ingelheim Investigational Site, Moscow
  - 1218.46.70004 Boehringer Ingelheim Investigational Site, Moscow
  - 1218.46.70006 Boehringer Ingelheim Investigational Site, Moscow
  - 1218.46.70008 Boehringer Ingelheim Investigational Site, Moscow
  - 1218.46.70005 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1218.46.70007 Boehringer Ingelheim Investigational Site, Saint Petersburg
- Sweden (5):
  - 1218.46.46002 Boehringer Ingelheim Investigational Site, Gothenburg
  - 1218.46.46004 Boehringer Ingelheim Investigational Site, Gothenburg
  - 1218.46.46003 Boehringer Ingelheim Investigational Site, Malmo
  - 1218.46.46005 Boehringer Ingelheim Investigational Site, Stockholm
  - 1218.46.46001 Boehringer Ingelheim Investigational Site, Uppsala
- Tunisia (5):
  - 1218.46.2162A Boehringer Ingelheim Investigational Site, Bab Sâadoun Tunis
  - 1218.46.2161A Boehringer Ingelheim Investigational Site, Tunis
  - 1218.46.2161B Boehringer Ingelheim Investigational Site, Tunis
  - 1218.46.2163A Boehringer Ingelheim Investigational Site, Tunis
  - 1218.46.2163B Boehringer Ingelheim Investigational Site, Tunis
- Ukraine (6):
  - 1218.46.38003 Boehringer Ingelheim Investigational Site, Kiev
  - 1218.46.38001 Boehringer Ingelheim Investigational Site, Lviv
  - 1218.46.38005 Boehringer Ingelheim Investigational Site, Lviv
  - 1218.46.38002 Boehringer Ingelheim Investigational Site, Odesa
  - 1218.46.38004 Boehringer Ingelheim Investigational Site, Odesa
  - 1218.46.38006 Boehringer Ingelheim Investigational Site, Vinnitsa

REFERENCES:
- [Derived] Lv Q, Shen J, Miao L, Ye B, Schepers C, Plat A, Shi Y. Early Combination Therapy with Linagliptin and Metformin in People with Type 2 Diabetes Improves Glycemic Control to HbA1c </= 6.5% without Increasing Hypoglycemia: Pooled Analysis of Two Randomized Clinical Trials. Diabetes Ther. 2020 Jun;11(6):1317-1330. doi: 10.1007/s13300-020-00819-9. Epub 2020 Apr 23. PMID 32328953

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Patients treated with matching placebo
- M500 Twice Daily (BID): Patients treated with Metformin 500 mg BID
- M1000 BID: Patients treated with Metformin 1000 mg BID
- Lina 5: Patients treated with Linagliptin 5 mg once daily (OD)
- L2.5+M500 BID: Patients treated with Linagliptin 2.5 mg + Metformin 500 mg BID
- L2.5 + M1000 BID: Patients treated with Linagliptin 2.5 mg + Metformin 1000 mg BID
- OL: L2.5+M1000 BID: Open label set: Linagliptin 2.5 mg + Metformin 1000 mg BID
Period: Overall Study
Arm/Group | Placebo | M500 Twice Daily (BID) | M1000 BID | Lina 5 | L2.5+M500 BID | L2.5 + M1000 BID | OL: L2.5+M1000 BID
Started | 72 | 144 | 147 | 142 | 143 | 143 | 66
Completed | 54 | 127 | 126 | 121 | 127 | 132 | 56
Not Completed | 18 | 17 | 21 | 21 | 16 | 11 | 10
Not completed — Adverse Event | 3 | 4 | 6 | 6 | 5 | 2 | 4
Not completed — Protocol Violation | 2 | 1 | 3 | 3 | 3 | 2 | 0
Not completed — Lost to Follow-up | 1 | 3 | 4 | 3 | 4 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 4 | 5 | 4 | 2 | 3 | 1
Not completed — Other reason (incl. lack of efficacy) | 7 | 5 | 3 | 5 | 2 | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- M500BID: Patients treated with Metformin 500mg BID
- M1000BID: Patients treated with Metformin 1000mg BID
- Lina5: Patients treated with Linagliptin 5mg OD
- L2.5+M500BID: Patients treated with Linagliptin 2.5mg+ Metformin 500mg BID
- L2.5+M1000BID: Patients treated with Linagliptin 2.5mg+ Metformin 1000mg BID
- L2.5+M1000BID (Open Label): Open label set: Linagliptin 2.5mg + Metformin 1000mg BID
- Total: Total of all reporting groups
Arm/Group | Placebo | M500BID | M1000BID | Lina5 | L2.5+M500BID | L2.5+M1000BID | L2.5+M1000BID (Open Label) | Total
Number analyzed (Participants) | 72 | 144 | 147 | 142 | 143 | 143 | 66 | 857
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.7 (11.0) | 52.9 (10.4) | 55.2 (10.6) | 56.2 (10.8) | 55.6 (11.2) | 56.4 (10.7) | 53.5 (11.1) | 55.2 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 62 | 69 | 62 | 70 | 66 | 40 | 405
  Male | 36 | 82 | 78 | 80 | 73 | 77 | 26 | 452
Body Mass Index (BMI) continuous [Mean (Standard Deviation); unit: kg/m^2] | 28.62 (5.17) | 28.92 (4.83) | 29.52 (5.31) | 28.95 (4.67) | 29.66 (5.31) | 28.55 (4.80) | 28.81 (4.93) | 29.07 (4.97)
Glycosylated Hemoglobin A1 (HbA1C) [Mean (Standard Deviation); unit: Percent] | 8.67 (0.95) | 8.66 (0.90) | 8.52 (0.87) | 8.70 (0.97) | 8.71 (0.95) | 8.68 (1.03) | 11.84 (1.42) | 8.91 (1.31)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] | 203.7 (51.2) | 191.2 (46.9) | 192.3 (52.8) | 195.3 (50.2) | 198.6 (60.2) | 196.9 (51.2) | 261.8 (80.9) | 200.2 (57.3)

OUTCOME MEASURES:

1. Primary Outcome: HbA1c Change From Baseline at Week 24
Description: HbA1c is measured as a percentage. Thus, this change from baseline reflects the Week 24 HbA1c percent minus the baseline HbA1c percent. Means are treatment adjusted for baseline HbA1c and previous anti-diabetic medication.
Time Frame: Baseline and week 24
Population: The Full Analysis Set (FAS) included all treated and randomised patients with a baseline and at least one on-treatment HbA1c measurement available. Last observation carried forward (LOCF) was used as the imputation rule.
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Placebo | M500BID | M1000BID | Lina5 | L2.5+M500BID | L2.5+M1000BID
Number analyzed (Participants) | 65 | 141 | 138 | 135 | 137 | 140
Percent | 0.13 (0.11) | -0.64 (0.08) | -1.07 (0.08) | -0.45 (0.08) | -1.22 (0.08) | -1.59 (0.08)
Statistical Analysis 1: Comparison: M500BID vs L2.5+M500BID; Metformin 500mg vs. Linagliptin 2.5mg with Metformin 500mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — hierarchical testing, no adjustment of p-values; Mean Difference (Final Values) = -0.58, 95% CI [-0.79 to -0.36], Standard Error of Mean 0.11
Statistical Analysis 2: Comparison: M1000BID vs L2.5+M1000BID; Metformin 1000mg vs. Linagliptin 2.5mg with Metformin 1000mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — hierarchical testing, no adjustment of p-values; Median Difference (Final Values) = -0.51, 95% CI [-0.73 to -0.30], Standard Error of Mean 0.11
Statistical Analysis 3: Comparison: Lina5 vs L2.5+M500BID; Linagliptin 5mg vs. Linagliptin 2.5mg with Metformin 500mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — hierarchical testing, no adjustment of p-values; Mean Difference (Final Values) = -0.77, 95% CI [-0.99 to -0.55], Standard Error of Mean 0.11
Statistical Analysis 4: Comparison: Lina5 vs L2.5+M1000BID; Linagliptin 5mg vs. Linagliptin 2.5mg with Metformin 1000mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — hierarchical testing, no adjustment of p-values; Mean Difference (Final Values) = -1.14, 95% CI [-1.36 to -0.92], Standard Error of Mean 0.11

2. Secondary Outcome: HbA1c Change From Baseline at Week 6
Description: HbA1c is measured as a percentage. Thus, this change from baseline reflects the Week 6 HbA1c percent minus the baseline HbA1c percent. Means are treatment adjusted for baseline HbA1c and previous anti-diabetic medication.
Time Frame: Baseline and week 6
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Placebo | M500BID | M1000BID | Lina5 | L2.5+M500BID | L2.5+M1000BID
Number analyzed (Participants) | 65 | 141 | 138 | 135 | 137 | 140
Percent | 0.03 (0.08) | -0.45 (0.05) | -0.61 (0.05) | -0.36 (0.06) | -0.86 (0.05) | -1.00 (0.05)
Statistical Analysis 1: Comparison: M500BID vs L2.5+M500BID; Metformin 500mg vs. Linagliptin 2.5mg with Metformin 500mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.41, 95% CI [-0.56 to -0.26], Standard Error of Mean 0.08
Statistical Analysis 2: Comparison: M1000BID vs L2.5+M1000BID; Metformin 1000mg vs. Linagliptin 2.5mg with Metformin 1000mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.38, 95% CI [-0.53 to -0.23], Standard Error of Mean 0.08
Statistical Analysis 3: Comparison: Lina5 vs L2.5+M500BID; Linagliptin 5mg vs Linagliptin 2.5mg with metformin 500mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.50, 95% CI [-0.65 to -0.35], Standard Error of Mean 0.08
Statistical Analysis 4: Comparison: Lina5 vs L2.5+M1000BID; Linagliptin 5mg vs. Linagliptin 2.5mg with Metformin 1000mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.64, 95% CI [-0.79 to -0.48], Standard Error of Mean 0.08

3. Secondary Outcome: HbA1c Change From Baseline at Week 12
Description: HbA1c is measured as a percentage. Thus, this change from baseline reflects the Week 12 HbA1c percent minus the baseline HbA1c percent. Means are treatment adjusted for baseline HbA1c and previous anti-diabetic medication.
Time Frame: Baseline and week 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Placebo | M500BID | M1000BID | Lina5 | L2.5+M500BID | L2.5+M1000BID
Number analyzed (Participants) | 65 | 141 | 138 | 135 | 137 | 140
Percent | 0.16 (0.11) | -0.61 (0.07) | -0.95 (0.07) | -0.42 (0.07) | -1.13 (0.07) | -1.37 (0.07)
Statistical Analysis 1: Comparison: M500BID vs L2.5+M500BID; Metformin 500mg vs. Linagliptin 2.5mg with Metformin 500mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.51, 95% CI [-0.72 to -0.31], Standard Error of Mean 0.10
Statistical Analysis 2: Comparison: M1000BID vs L2.5+M1000BID; Metformin 1000mg vs. Linagliptin 2.5mg with Metformin 1000mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.42, 95% CI [-0.63 to -0.22], Standard Error of Mean 0.10
Statistical Analysis 3: Comparison: Lina5 vs L2.5+M500BID; Linagliptin 5mg vs. Linagliptin 2.5mg with Metformin 500mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.71, 95% CI [-0.92 to -0.51], Standard Error of Mean 0.11
Statistical Analysis 4: Comparison: Lina5 vs L2.5+M1000BID; Linagliptin 5mg vs. Linagliptin 2.5mg with Metformin 1000mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.95, 95% CI [-1.16 to -0.75], Standard Error of Mean 0.10

4. Secondary Outcome: HbA1c Change From Baseline at Week 18
Description: HbA1c is measured as a percentage. Thus, this change from baseline reflects the Week 18 HbA1c percent minus the baseline HbA1c percent. Means are treatment adjusted for baseline HbA1c and previous anti-diabetic medication.
Time Frame: Baseline and week 18
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Placebo | M500BID | M1000BID | Lina5 | L2.5+M500BID | L2.5+M1000BID
Number analyzed (Participants) | 65 | 141 | 138 | 135 | 137 | 140
Percent | 0.16 (0.12) | -0.66 (0.08) | -1.06 (0.08) | -0.45 (0.08) | -1.17 (0.08) | -1.54 (0.08)
Statistical Analysis 1: Comparison: M500BID vs L2.5+M500BID; Metformin 500mg vs. Linagliptin 2.5mg with Metformin 500mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.51, 95% CI [-0.73 to -0.29], Standard Error of Mean 0.11
Statistical Analysis 2: Comparison: M1000BID vs L2.5+M1000BID; Metformin 1000mg vs. Linagliptin 2.5mg with Metformin 1000mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.47, 95% CI [-0.69 to -0.26], Standard Error of Mean 0.11
Statistical Analysis 3: Comparison: Lina5 vs L2.5+M500BID; Linagliptin 5mg vs. Linagliptin 2.5mg with Metformin 500mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.72, 95% CI [-0.94 to -0.49], Standard Error of Mean 0.11
Statistical Analysis 4: Comparison: Lina5 vs L2.5+M1000BID; Linagliptin 5mg vs. Linagliptin 2.5mg with Metformin 1000mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -1.08, 95% CI [-1.30 to -0.86], Standard Error of Mean 0.11

5. Secondary Outcome: FPG Change From Baseline at Week 24
Description: This change from baseline reflects the Week 24 FPG minus the baseline FPG. Means are treatment adjusted for baseline HbA1c, baseline FPG and previous anti-diabetic medication.
Time Frame: Baseline and week 24
Population: This population includes the FAS using the LOCF imputation, with the further restriction of patients with a baseline and post-baseline FPG value.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | M500BID | M1000BID | Lina5 | L2.5+M500BID | L2.5+M1000BID
Number analyzed (Participants) | 61 | 136 | 132 | 134 | 135 | 136
mg/dL | 10.2 (5.3) | -15.8 (3.5) | -32.2 (3.6) | -8.6 (3.6) | -33.2 (3.5) | -49.4 (3.5)
Statistical Analysis 1: Comparison: M500BID vs L2.5+M500BID; Metformin 500mg vs. Linagliptin 2.5mg with Metformin 500mg; Test type: Superiority or Other; p = 0.0005, ANCOVA; Mean Difference (Final Values) = -17.4, 95% CI [-27.2 to -7.6], Standard Error of Mean 5.0
Statistical Analysis 2: Comparison: M1000BID vs L2.5+M1000BID; Metformin 1000mg vs. Linagliptin 2.5mg with Metformin 1000mg; Test type: Superiority or Other; p = 0.0006, ANCOVA; Mean Difference (Final Values) = -17.2, 95% CI [-27.1 to -7.3], Standard Error of Mean 5.0
Statistical Analysis 3: Comparison: Lina5 vs L2.5+M500BID; Linagliptin 5mg vs. Linagliptin 2.5mg with Metformin 500mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -24.6, 95% CI [-34.4 to -14.8], Standard Error of Mean 5.0
Statistical Analysis 4: Comparison: Lina5 vs L2.5+M1000BID; Linagliptin 5mg vs. linagliptin 2.5mg with metformin 1000mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -40.8, 95% CI [-50.6 to -31.0], Standard Error of Mean 5.0

6. Secondary Outcome: FPG Change From Baseline at Week 2
Description: This change from baseline reflects the Week 2 FPG minus the baseline FPG. Means are treatment adjusted for baseline HbA1c, baseline FPG and previous anti-diabetic medication.
Time Frame: Baseline and week 2
Population: as for outcome 5
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | M500BID | M1000BID | Lina5 | L2.5+M500BID | L2.5+M1000BID
Number analyzed (Participants) | 61 | 136 | 132 | 134 | 135 | 136
mg/dL | 5.3 (4.3) | -19.6 (2.9) | -21.8 (2.9) | -13.0 (2.9) | -34.5 (2.9) | -38.6 (2.9)
Statistical Analysis 1: Comparison: M500BID vs L2.5+M500BID; Metformin 500mg vs. Linagliptin 2.5mg with Metformin 500mg; Test type: Superiority or Other; p = 0.0003, ANCOVA; Mean Difference (Final Values) = -14.9, 95% CI [-22.9 to -6.8], Standard Error of Mean 4.1
Statistical Analysis 2: Comparison: M1000BID vs L2.5+M1000BID; Metformin 1000mg vs. Linagliptin 2.5mg with Metformin 1000mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -16.8, 95% CI [-24.9 to -8.8], Standard Error of Mean 4.1
Statistical Analysis 3: Comparison: Lina5 vs L2.5+M500BID; Linagliptin 5mg vs. Linagliptin 2.5mg with Metformin 500mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -21.5, 95% CI [-29.5 to -13.4], Standard Error of Mean 4.1
Statistical Analysis 4: Comparison: Lina5 vs L2.5+M1000BID; Linagliptin 5mg vs. Linagliptin 2.5mg with Metformin 1000mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -25.6, 95% CI [-33.6 to -17.6], Standard Error of Mean 4.1

7. Secondary Outcome: FPG Change From Baseline at Week 6
Description: This change from baseline reflects the Week 6 FPG minus the baseline FPG. Means are treatment adjusted for baseline HbA1c, baseline FPG and previous anti-diabetic medication.
Time Frame: Baseline and week 6
Population: as for outcome 5
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | M500BID | M1000BID | Lina5 | L2.5+M500BID | L2.5+M1000BID
Number analyzed (Participants) | 61 | 136 | 132 | 134 | 135 | 136
mg/dL | 6.2 (4.7) | -20.8 (3.2) | -31.6 (3.2) | -10.8 (3.2) | -38.7 (3.2) | -48.3 (3.2)
Statistical Analysis 1: Comparison: M500BID vs L2.5+M500BID; Metformin 500mg vs. Linagliptin 2.5mg with Metformin 500mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -17.9, 95% CI [-26.7 to -9.1], Standard Error of Mean 4.5
Statistical Analysis 2: Comparison: M1000BID vs L2.5+M1000BID; Metformin 1000mg vs. Linagliptin 2.5mg with Metformin 1000mg; Test type: Superiority or Other; p = 0.0002, ANCOVA; Mean Difference (Final Values) = -16.8, 95% CI [-25.6 to -7.9], Standard Error of Mean 4.5
Statistical Analysis 3: Comparison: Lina5 vs L2.5+M500BID; Linagliptin 5mg vs. Linagliptin 2.5mg with Metformin 500mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -27.9, 95% CI [-36.7 to -19.1], Standard Error of Mean 4.5
Statistical Analysis 4: Comparison: Lina5 vs L2.5+M1000BID; Linagliptin 5mg vs. Linagliptin 2.5mg with Metformin 1000mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -37.6, 95% CI [-46.4 to -28.8], Standard Error of Mean 4.5

8. Secondary Outcome: FPG Change From Baseline at Week 12
Description: This change from baseline reflects the Week 12 FPG minus the baseline FPG. Means are treatment adjusted for baseline HbA1c, baseline FPG and previous anti-diabetic medication.
Time Frame: Baseline and week 12
Population: as for outcome 5
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | M500BID | M1000BID | Lina5 | L2.5+M500BID | L2.5+M1000BID
Number analyzed (Participants) | 61 | 136 | 132 | 134 | 135 | 136
mg/dL | 8.9 (5.0) | -21.8 (3.3) | -31.9 (3.4) | -8.4 (3.4) | -36.2 (3.4) | -49.9 (3.3)
Statistical Analysis 1: Comparison: M500BID vs L2.5+M500BID; Metformin 500mg vs. Linagliptin 2.5mg with Metformin 500mg; Test type: Superiority or Other; p = 0.0024, ANCOVA; Mean Difference (Final Values) = -14.4, 95% CI [-23.7 to -5.1], Standard Error of Mean 4.7
Statistical Analysis 2: Comparison: M1000BID vs L2.5+M1000BID; Metformin 1000mg vs. Linagliptin 2.5mg with Metformin 1000mg; Test type: Superiority or Other; p = 0.0002, ANCOVA; Mean Difference (Final Values) = -18.0, 95% CI [-27.4 to -8.7], Standard Error of Mean 4.8
Statistical Analysis 3: Comparison: Lina5 vs L2.5+M500BID; Linagliptin 5mg vs. Linagliptin 2.5mg with Metformin 500mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -27.8, 95% CI [-37.1 to -18.5], Standard Error of Mean 4.7
Statistical Analysis 4: Comparison: Lina5 vs L2.5+M1000BID; Linagliptin 5mg vs. Linagliptin 2.5mg with Metformin 1000mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -41.5, 95% CI [-50.8 to -32.2], Standard Error of Mean 4.7

9. Secondary Outcome: FPG Change From Baseline at Week 18
Description: This change from baseline reflects the Week 18 FPG minus the baseline FPG. Means are treatment adjusted for baseline HbA1c, baseline FPG and previous anti-diabetic medication.
Time Frame: Baseline and week 18
Population: as for outcome 5
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | M500BID | M1000BID | Lina5 | L2.5+M500BID | L2.5+M1000BID
Number analyzed (Participants) | 61 | 136 | 132 | 134 | 135 | 136
mg/dL | 7.3 (5.1) | -13.7 (3.4) | -30.3 (3.5) | -9.2 (3.4) | -34.6 (3.4) | -48.1 (3.4)
Statistical Analysis 1: Comparison: M500BID vs L2.5+M500BID; Metformin 500mg vs. Linagliptin 2.5mg with Metformin 500mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -20.9, 95% CI [-30.4 to -11.4], Standard Error of Mean 4.8
Statistical Analysis 2: Comparison: M1000BID vs L2.5+M1000BID; Metformin 1000mg vs. Linagliptin 2.5mg with Metformin 1000mg; Test type: Superiority or Other; p = 0.0003, ANCOVA; Mean Difference (Final Values) = -17.9, 95% CI [-27.4 to -8.3], Standard Error of Mean 4.9
Statistical Analysis 3: Comparison: Lina5 vs L2.5+M500BID; Linagliptin 5mg vs. Linagliptin 2.5mg with Metformin 500mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -25.4, 95% CI [-35.0 to -15.9], Standard Error of Mean 4.9
Statistical Analysis 4: Comparison: Lina5 vs L2.5+M1000BID; Linagliptin 5 mg vs. Linagliptin 2.5 mg with Metformin 1000 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -39.0, 95% CI [-48.5 to -29.4], Standard Error of Mean 4.9

10. Secondary Outcome: Percentage of Patients With HbA1c <7.0% at Week 24
Description: The percentage of patients with an HbA1c value below 7% at week 24 was calculated for each treatment arm. If a patient did not have an HbA1c value at week 24 they were considered a failure, so HbA1c above 7%.
Time Frame: Baseline and Week 24
Population: FAS treated and randomised patients with baseline HbA1c >= 7.0%. Non-completers were considered as failure imputation (NCF).
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | M500BID | M1000BID | Lina5 | L2.5+M500BID | L2.5+M1000BID
Number analyzed (Participants) | 65 | 140 | 137 | 135 | 136 | 138
percentage of patients | 10.8 (0) | 18.6 (0) | 30.7 (0) | 10.4 (0) | 30.1 (0) | 53.6 (0)
Statistical Analysis 1: Comparison: M500BID vs L2.5+M500BID; Metformin 500mg vs. Linagliptin 2.5mg with Metformin 500mg; Test type: Superiority or Other; p = 0.0062, Regression, Logistic; The odds-ratio is based on a logistic regression model including baseline HbA1c and previous antidiabetic medication; Odds Ratio (OR) = 2.372, 95% CI [1.278 to 4.402]
Statistical Analysis 2: Comparison: M1000BID vs L2.5+M1000BID; Metformin 1000mg vs. Linagliptin 2.5mg with Metformin 1000mg; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; The odds-ratio is based on a logistic regression model including baseline HbA1c and previous antidiabetic medication; Odds Ratio (OR) = 4.163, 95% CI [2.343 to 7.397]
Statistical Analysis 3: Comparison: Lina5 vs L2.5+M500BID; Linagliptin 5mg vs. Linagliptin 2.5mg with Metformin 500mg; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; The odds-ratio is based on a logistic regression model including baseline HbA1c and previous antidiabetic medication; Odds Ratio (OR) = 4.854, 95% CI [2.363 to 9.973]
Statistical Analysis 4: Comparison: Lina5 vs L2.5+M1000BID; Linagliptin 5mg vs. Linagliptin 2.5mg with Metformin 1000mg; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; The odds-ratio is based on a logistic regression model including baseline HbA1c and previous antidiabetic medication; Odds Ratio (OR) = 17.094, 95% CI [8.238 to 35.471]

11. Secondary Outcome: Percentage of Patients With HbA1c<7.0 at Week 24
Description: as for outcome 10
Time Frame: Baseline and Week 24
Population: The FAS included all treated and randomised patients with a baseline and at least one on-treatment HbA1c measurement available. Non-completers were considered as failure imputation (NCF).
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | M500BID | M1000BID | Lina5 | L2.5+M500BID | L2.5+M1000BID
Number analyzed (Participants) | 65 | 141 | 138 | 135 | 137 | 140
percentage of patients | 10.8 | 19.1 | 31.2 | 10.4 | 30.7 | 54.3

12. Secondary Outcome: Percentage of Patients With HbA1c <6.5% at Week 24
Description: The percentage of patients with an HbA1c value below 6.5% at week 24 was calculated for each treatment arm. If a patient did not have an HbA1c value at week 24 they were considered a failure, so HbA1c above 6.5%. Only patients with baseline HbA1c =< 6.5%
Time Frame: Baseline and Week 24
Population: FAS treated and randomised patients with baseline HbA1c >= 6.5%. Non-completers were considered as failure imputation (NCF).
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | M500BID | M1000BID | Lina5 | L2.5+M500BID | L2.5+M1000BID
Number analyzed (Participants) | 65 | 141 | 138 | 135 | 137 | 140
percentage of patients | 3.1 (0) | 5.0 (0) | 12.3 (0) | 3.7 (0) | 13.1 (0) | 27.1 (0)
Statistical Analysis 1: Comparison: M500BID vs L2.5+M500BID; Metformin 500mg vs. Linagliptin 2.5mg with Metformin 500mg; Test type: Superiority or Other; p = 0.0102, Regression, Logistic; The odds-ratio is based on a logistic regression model including baseline HbA1c and previous antidiabetic medication; Odds Ratio (OR) = 3.465, 95% CI [1.342 to 8.943]
Statistical Analysis 2: Comparison: M1000BID vs L2.5+M1000BID; Metformin 1000mg vs. Linagliptin 2.5mg with Metformin 1000mg; Test type: Superiority or Other; p = 0.0004, Regression, Logistic; The odds-ratio is based on a logistic regression model including baseline HbA1c and previous antidiabetic medication; Odds Ratio (OR) = 3.521, 95% CI [1.747 to 7.094]
Statistical Analysis 3: Comparison: Lina5 vs L2.5+M500BID; Linagliptin 5mg vs. Linagliptin 2.5mg with Metformin 500mg; Test type: Superiority or Other; p = 0.0053, Regression, Logistic; The odds-ratio is based on a logistic regression model including baseline HbA1c and previous antidiabetic medication; Odds Ratio (OR) = 4.521, 95% CI [1.564 to 13.069]
Statistical Analysis 4: Comparison: Lina5 vs L2.5+M1000BID; Linagliptin 5mg vs. Linagliptin 2.5mg with Metformin 1000mg; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; The odds-ratio is based on a logistic regression model including baseline HbA1c and previous antidiabetic medication; Odds Ratio (OR) = 11.947, 95% CI [4.314 to 33.080]

13. Secondary Outcome: Percentage of Patients With HbA1c < 6.5% at Week 24
Description: The percentage of patients with an HbA1c value below 6.5% at week 24 was calculated for each treatment arm. If a patient did not have an HbA1c value at week 24 they were considered a failure, so HbA1c above 6.5%
Time Frame: Baseline and Week 24
Population: as for outcome 11
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | M500BID | M1000BID | Lina5 | L2.5+M500BID | L2.5+M1000BID
Number analyzed (Participants) | 65 | 141 | 138 | 135 | 137 | 140
percentage of patients | 3.1 | 5.0 | 12.3 | 3.7 | 13.1 | 27.1

14. Secondary Outcome: Percentage of Patients With HbA1c Lowering by 0.5% at Week 24
Description: The percentage of patients with an HbA1c reduction from baseline greater than 0.5% at week 24 was calculated for each treatment arm. If a patient did not have an HbA1c value at week 24 they were considered a failure, so HbA1c reduction less than 0.5%.
Time Frame: Baseline and week 24
Population: as for outcome 11
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | M500BID | M1000BID | Lina5 | L2.5+M500BID | L2.5+M1000BID
Number analyzed (Participants) | 65 | 141 | 138 | 135 | 137 | 140
percentage of patients | 29.2 (0) | 46.1 (0) | 65.9 (0) | 42.2 (0) | 71.5 (0) | 81.4 (0)
Statistical Analysis 1: Comparison: M500BID vs L2.5+M500BID; Metformin 500mg vs. Linagliptin 2.5mg with Metformin 500mg; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; The odds-ratio is based on a logistic regression model including baseline HbA1c and previous antidiabetic medication; Odds Ratio (OR) = 3.181, 95% CI [1.903 to 5.316]
Statistical Analysis 2: Comparison: M1000BID vs L2.5+M1000BID; Metformin 1000mg vs. Linagliptin 2.5mg with Metformin 1000mg; Test type: Superiority or Other; p = 0.0027, Regression, Logistic; The odds-ratio is based on a logistic regression model including baseline HbA1c and previous antidiabetic medication; Odds Ratio (OR) = 2.382, 95% CI [1.352 to 4.196]
Statistical Analysis 3: Comparison: Lina5 vs L2.5+M500BID; Linagliptin 5mg vs. Linagliptin 2.5mg with Metformin 500mg; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; The odds-ratio is based on a logistic regression model including baseline HbA1c and previous antidiabetic medication; Odds Ratio (OR) = 3.622, 95% CI [2.153 to 6.093]
Statistical Analysis 4: Comparison: Lina5 vs L2.5+M1000BID; Linagliptin 5mg vs. Linagliptin 2.5mg with Metformin 1000mg; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; The odds-ratio is based on a logistic regression model including baseline HbA1c and previous antidiabetic medication; Odds Ratio (OR) = 6.529, 95% CI [3.724 to 11.445]

15. Secondary Outcome: Adjusted Means for 2h Post-Prandial Glucose (PPG) Change From Baseline at Week 24
Description: This change from baseline reflects the Week 24 2h PPG minus the baseline 2h PPG. Means are treatment adjusted for baseline HbA1c, baseline 2h PPG and previous anti-diabetic medication.
Time Frame: Baseline and week 24
Population: Meal tolerance test (MTT) set (patients with adequate MTT results available at the beginning and end of the randomised treatment period)
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | M500BID | M1000BID | Lina5 | L2.5+M500BID | L2.5+M1000BID
Number analyzed (Participants) | 6 | 15 | 14 | 12 | 10 | 12
mg/dL | -35.4 (23.2) | -82.9 (14.4) | -87.2 (14.8) | -35.3 (16.1) | -86.0 (17.5) | -109.2 (16.2)
Statistical Analysis 1: Comparison: M500BID vs L2.5+M500BID; Metformin 500mg vs. Linagliptin 2.5mg with Metformin 500mg; Test type: Superiority or Other; p = 0.8893, ANCOVA; Mean Difference (Final Values) = -3.2, 95% CI [-48.5 to 42.2], Standard Error of Mean 22.7
Statistical Analysis 2: Comparison: M1000BID vs L2.5+M1000BID; Metformin 1000mg vs. Linagliptin 2.5mg with Metformin 1000mg; Test type: Superiority or Other; p = 0.3234, ANCOVA; Mean Difference (Final Values) = -22.0, 95% CI [-66.2 to 22.2], Standard Error of Mean 22.1
Statistical Analysis 3: Comparison: Lina5 vs L2.5+M500BID; Linagliptin 5mg vs. Linagliptin 2.5mg with Metformin 500mg; Test type: Superiority or Other; p = 0.0373, ANCOVA; Mean Difference (Final Values) = -50.8, 95% CI [-98.5 to -3.1], Standard Error of Mean 23.8
Statistical Analysis 4: Comparison: Lina5 vs L2.5+M1000BID; Linagliptin 5mg vs. Linagliptin 2.5mg with Metformin 1000mg; Test type: Superiority or Other; p = 0.0018, ANCOVA; Mean Difference (Final Values) = -73.9, 95% CI [-119.3 to -28.6], Standard Error of Mean 22.7

16. Secondary Outcome: HbA1c Change From Baseline at Week 24 for Open-label Patients
Description: HbA1c is measured as a percentage. Thus, this change from baseline reflects the Week 24 HbA1c percent minus the baseline HbA1c percentage. Mean is unadjusted.
Time Frame: Baseline and week 24
Population: The open label set (OLS) included all patients with baseline HbA1c too high to be randomised and were assigned open-label medication, also with an on treatment HbA1c value. The Open label Set (OLS) included all patients treated with at least one dose on open-label L2.5+M1000 medication.
Measure: Mean (Standard Deviation); unit: Percent
Groups:
- OL: L2.5+M1000BID: Open label set: Linagliptin 2.5mg + Metformin 1000mg twice daily (BID)
Arm/Group | OL: L2.5+M1000BID
Number analyzed (Participants) | 65
Percent | -3.19 (2.04)

17. Secondary Outcome: FPG Change From Baseline at Week 24 for Open-label Patients
Description: This change from baseline reflects the Week 24 FPG minus the baseline FPG. Mean is unadjusted.
Time Frame: Baseline and week 24
Population: The open label set (OLS) included all patients with baseline HbA1c too high to be randomised and were assigned open-label medication, also with a baseline on treatment HbA1c value. The Open label Set (OLS) included all patients treated with at least one dose on open-label L2.5+M1000 medication.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | OL: L2.5+M1000BID
Number analyzed (Participants) | 55
mg/dL | -73.58 (70.94)

18. Secondary Outcome: Use of Rescue Therapy
Description: The use of rescue therapy (SUs, thiazolidinediones [TZDs], or insulin) was permitted only during the randomised treatment period of the trial (i.e. Visits 3 to 7), and was to be administered only if a patient had a 'confirmed' glucose level after an overnight fast.
Time Frame: 24 weeks
Population: Percentage of patients requiring rescue therapy
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | M500BID | M1000BID | Lina5 | L2.5+M500BID | L2.5+M1000BID
Number analyzed (Participants) | 65 | 141 | 138 | 135 | 137 | 140
percentage of participants | 29.2 | 13.5 | 8.0 | 11.1 | 7.3 | 4.3
Statistical Analysis 1: Comparison: M1000BID vs L2.5+M1000BID; Test type: Superiority or Other; p = 0.0445, Regression, Logistic; Odds Ratio (OR) = 0.326, 95% CI 2-sided [0.109 to 0.973]
Statistical Analysis 2: Comparison: Lina5 vs L2.5+M1000BID; Test type: Superiority or Other; p = 0.0151, Regression, Logistic; Odds Ratio (OR) = 0.274, 95% CI 2-sided [0.096 to 0.779]
Statistical Analysis 3: Comparison: M500BID vs L2.5+M500BID; Test type: Superiority or Other; p = 0.0490, Regression, Logistic; Odds Ratio (OR) = 0.420, 95% CI 2-sided [0.177 to 0.996]
Statistical Analysis 4: Comparison: Lina5 vs L2.5+M500BID; Test type: Superiority or Other; p = 0.2617, Regression, Logistic; Odds Ratio (OR) = 0.598, 95% CI 2-sided [0.244 to 1.467]

ADVERSE EVENTS:
Time Frame: Day of first dose until day of last dose plus 7 days
Groups:
- M500 BID: Patients treated with Metformin 500 mg BID
- M1000 BID: Patients treated with Metformin 1000 mg bis in die (BID)
- L2.5+M500 BID: Patients treated with Linagliptin 2.5 mg + Metformin 500 mg bis in die (BID)
- L2.5 + M1000 BID: Patients treated with Linagliptin 2.5 mg + Metformin 1000 mg bis in die (BID)
- OL: L2.5+M1000 BID: Open label set: Linagliptin 2.5 mg + Metformin 1000 mg bis in die (BID)
Arm/Group | Placebo | M500 BID | M1000 BID | Lina 5 | L2.5+M500 BID | L2.5 + M1000 BID | OL: L2.5+M1000 BID
Serious Adverse Events (participants affected / at risk) | 1/72 | 3/144 | 6/147 | 3/142 | 2/143 | 2/143 | 1/66
Other Adverse Events (participants affected / at risk) | 20/72 | 27/144 | 27/147 | 31/142 | 31/143 | 36/143 | 18/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=72) | M500 BID (N=144) | M1000 BID (N=147) | Lina 5 (N=142) | L2.5+M500 BID (N=143) | L2.5 + M1000 BID (N=143) | OL: L2.5+M1000 BID (N=66)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Left ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hyperparathyroidism primary (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malaria (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Plasmodium falciparum infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Breast cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abortion induced (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=72) | M500 BID (N=144) | M1000 BID (N=147) | Lina 5 (N=142) | L2.5+M500 BID (N=143) | L2.5 + M1000 BID (N=143) | OL: L2.5+M1000 BID (N=66)
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 8 | 5 | 7 | 11 | 4
Nasopharyngitis (Infections and infestations) | 1 | 4 | 4 | 8 | 12 | 6 | 2
Glomerular filtration rate decreased (Investigations) | 4 | 4 | 3 | 5 | 2 | 6 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 10 | 11 | 3 | 5 | 5 | 2 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 5 | 5 | 2 | 8 | 2
Hypertension (Vascular disorders) | 4 | 5 | 4 | 3 | 5 | 5 | 3
Urinary tract infection (Infections and infestations) | 2 | 3 | 3 | 2 | 2 | 7 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.